CLINICAL TRIAL: NCT03622190
Title: A Longitudinal Investigation of the Factors Associated With Increased Risk of Playing-related Musculoskeletal Disorders Among Music Students
Brief Title: The RISMUS Cohort Study: Risk Among Music Students.
Acronym: RISMUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Cinzia Cruder, Principal Investigator, Queen Margaret University
Other Study IDs: REP 0177
Record Dates: First submitted 2018-07-31; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Upper Limb Injury
Keywords: playing-related musculoskeletal disorder (PRMD); music students; pain; musculoskeletal (MSK) disorder
MeSH Terms: conditions — Arm Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Music students who are free of pain, PRMDs and/or MSK problems at baseline data collection
- Cohort 2: Music students who aren't free of pain, PRMDs and/or MSK problems at baseline data collection

SUMMARY:
This observational cohort study involves repeated cross-sectional observations in order to identify those factors associated with increased risk of PRMDs among music students.

All pre-college and university-level students from several European music academies will receive an invitation to complete a web-based questionnaire survey at each of three occasions (baseline; 6-months follow-up; 12-months follow-up).

DETAILED DESCRIPTION:
Professional musicians are exposed to chronic high volume of continuous and repeated physical movements, sometimes in challenging and ergonomically unfavourable anatomical body positions, in order to acquire and improve technical playing skills. As a consequence, musicians are vulnerable to developing adverse playing-related musculoskeletal disorders (PRMDs) that may affect the manner in which and the extent to which music can be practised and performed.

In order to find out effective solutions for PRMDs and to develop future preventive measures, it is fundamental to firstly identify the main risk factors that play a significant role in the development of adverse musculoskeletal (MSK) conditions and symptoms.

The longitudinal cohort study will be conducted through the following three phases:

1. a baseline cross-sectional survey (i.e. web-based questionnaire) to characterise the study population and subgroups, and form the basis for the evaluation of associated factors and relationships with the development of PRMDs;
2. a 6-months follow-up survey, and
3. a 12-months follow-up survey.

After the first baseline data collection (Phase 1), the cohort of students will be broken down into:

* Cohort 1: music students (both pre-college and university-level) who are free of pain and PRMDs at baseline data collection
* Cohort 2: music students (both pre-college and university-level) who aren't free of pain and PRMDs at baseline data collection

Afterwards, the two cohorts will be followed and invited for reassessment at 6 months (Phase 2) and 12 months (Phase 3).

Both the follow-ups will permit longitudinal change in outcome scores to be generated and compared (longitudinal comparisons) for strength and progression of association, alongside those from absolute outcome scores at several cross-sectional analyses.

The web-based survey will include questions about any pain, PRMD and/or MSK problem they may have due to their musical practice, and different outcome measures (i.e. lifestyle and physical activity, practice habits, behaviour toward prevention and health history, level of stress, perfectionism, fatigue and disability).

The outcome measures have been selected according to the relevant findings of previous cross-sectional studies and systematic reviews among the performing arts literature.

Each outcome measure correspond to a suspected factor that may be associated with the development of a PRMD.

To the best of our knowledge, no other longitudinal studies on risk factors for PRMDs have been conducted so far. Therefore, the study can be considered as an opportunity to fill the gaps of current research on PRMDs and generate new knowledge in educational and employment musical contexts.

ELIGIBILITY:
Inclusion Criteria:

* All pre-college and university-level students from music academies, with a classical instrument as main subject.

Exclusion Criteria:

* Music students without a classical instrument as main subject (composers and conductors)
* Positive history for neurological, rheumatic, psychological disorders or emotional distress, as well as surgery of the upper limbs and/or the spine in the last 12 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pre-college and university-level students from ten music academies, with a classical instrument as main subject (composers and conductors will be excluded) will receive an invitation to complete a web-based questionnaire survey.
  Pre-college will include third-year and fourth-year students (age: 18 and 19 years old). University-level will include students enrolled in the first, second and third year of the Bachelor degree course (age: between 19, 20 and 22, 23 years old), as well as students enrolled in the first, second and third year of Master degree course (age: between 22, 23 and 35 years old).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Presence of pain or musculoskeletal (MSK) disorder | up to 12 months
  The presence of pain and/or MSK problems will be assessed through the following question: "When did you last experience a bout of significant pain and/or musculoskeletal problem?"
Presence of playing-related musculoskeletal disorders (PRMDs) | one month
  Self reported PRMDs according to the definition: "any pain and/or musculoskeletal problem interfered with students' ability to play their musical instrument at the level to which they are accustomed"
Severity of pain or MSK disorder | one month
  Respondents are asked to assign a number, from zero (no pain) to ten (the worst possible pain), to the severity of their pain.
Location of pain | one month
  Respondents are asked to indicate where they have pain and/or MSK disorders by clicking on the part(s) in which they have or have had their pain and/or MSK problem during the last month.
Pain Disability Index | one month
  A short, self-report instrument for measuring the degree of interference with normal role functioning caused by pain. The respondent uses an 11-point scale ranging from 0 (no disability) to 10 (total disability) to rate the degree to which pain interferes with functioning in the following seven areas: family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity. The total score can range from 0 to 70.to participate in essential life activities.
A 2-item short form of the Pain Self-efficacy Questionnaire (PSEQ-2) | one month
  Respondents are asked to rate how confidently they can perform work and normal life activities, despite their pain. They answer by circling a number on a 7-point Likert scale under each item, where 0 = not at all confident and 6= completely confident in the last month.
Quick Dash - Performing Arts Section | one week
  This questions relate to the impact of your pain on playing students' practice. Respondents rate each item based on their experience over the preceding week on a 5-point Likert-type scale, increasing from 1 to 5 in level of difficulty/severity.
Self-rated health (SRH) | 12 months
  The SHR is a simple measure which is usually assessed as a single-item: "In general, would you say your health is", with the response items "excellent," "very good," "good," "fair," or "poor" to assess health status.

SECONDARY OUTCOMES:
Standardised Nordic Questionnaire (SNQ) | 12 months
  A general questionnaire on 12-months prevalence of troubles in nine symptom sites being neck, shoulders, upper back, elbows, low back, wrist/hands, hips/thighs, knees and ankles/feet.
Internation Physical Activity Questionnaire - short form (IPAQ-SF) | one week
  IPAQ-SF investigates the physical activity of four intensity levels (i.e. vigorous-intensity activity, moderate-intensity activity, walking, and sitting) in the past week.
Kessler Psychological Distress Scale (K10) | four weeks
  A brief measure of non-specific psychological distress in the anxiety-depression spectrum. The K10 comprises ten questions about psychological distress designed to measure anxiety and depression. Each question is related to a specific emotional state and each has a five-level response scale. It is designed to quantify the frequency and severity of anxiety- and depression-related symptoms experienced in the past four weeks.
Multidimensional Perfectionism Scale - short form (HFMPS-SF) | 12 months
  The HFMPS-SF is a 15-item questionnaire to measure trait perfectionism. Respondents rate each item on a 7-point Likert scale, increasing in level of agreement (from 1 "disagree" to 7 "agree"). Items are structured according to three subscales: self-oriented (SOP), other-oriented (OOP), and socially prescribed perfectionism (SPP), where higher scores on each scale, indicating higher levels of perfectionistic attitudes and behaviours.
The Chalder Fatigue Scale (CFQ-11) | one month
  The CFQ-11 is a reliable measure (Cronbach α = 0.90) to assess the severity of tiredness among population (Chalder et al. 1993). Each of the eleven items are answered on a 4-point Likert-type, from 1 (asymptomatic) increasing to 4 as responses become more symptomatic. The respondent's global score can range from 0 to 33, where higher scores indicate greater tiredness. The global score also includes two dimensions-physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11).

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Cruder, MA, Principal Investigator — Queen Margaret University

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available. Even if made available, individual participant's information obtained as a result of this research project will be considered confidential and disclosure to third parties will be prohibited (unless required by law). It will only be the clinical information that will be shared.

REFERENCES:
- [Derived] Cruder C, Koufaki P, Barbero M, Gleeson N. A longitudinal investigation of the factors associated with increased RISk of playing-related musculoskeletal disorders in MUsic students (RISMUS): a study protocol. BMC Musculoskelet Disord. 2019 Feb 8;20(1):64. doi: 10.1186/s12891-019-2440-4. PMID 30736779

DOCUMENTS (1):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03622190/Prot_000.pdf